CLINICAL TRIAL: NCT00888043
Title: A Phase I/Biomarker Study of Bevacizumab in Combination With CNTO 95 in Patients With Refractory Solid Tumors
Brief Title: Safety/Biomarker Study of CNTO 95 and Avastin in Solid Tumors
Acronym: CNTO95/Avastin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: Centocor, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00004929
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Solid Tumors
Keywords: solid tumors; avastin; Phase I; combination therapy; bevacizumab
MeSH Terms: interventions — intetumumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): CNTO 95 and avastin
  Interventions: Drug: CNTO 95 and avastin

INTERVENTIONS:
Drug: CNTO 95 and avastin — STAGE 1 (Dose escalation) Cohort # subjects CNTO 95 Bevacizumab
  * 2 3-6 2.5 mg/kg IV Q3 weeks 7.5 mg/kg IV Q3 weeks
  * 1 3-6 2.5 mg/kg IV Q3 weeks 15 mg/kg IV Q3 weeks
    1. 3-6 5 mg/kg IV Q3weeks 15 mg/kg IV Q3 weeks
    2. 3-6 10 mg/kg IV Q3 weeks 15 mg/kg IV Q3 weeks STAGE 2 (Biomarker) Cohort # subjects CNTO 95 Bevacizumab
    3. 20 Recommended Phase II Dose Recommended Phase II Dose
  Other Names: bevacizumab

SUMMARY:
The purpose of this research study is to find out what side effects the combination of the two study drugs, bevacizumab (Avastin) and CNTO 95 have on the body and to determine the highest dose of CNTO 95 that can be given with bevacizumab that is safe and well tolerated.

DETAILED DESCRIPTION:
Targeting molecular pathways of tumor growth has recently become a major focus of anti-cancer treatments. The VEGF pathway has demonstrated significant mitogenic activity for arterial, venous, and lymphatic endothelial cells, induction of vascular permeability for extracellular remodeling, and activity as an endothelial cell growth factor. The proof of principle that targeting the VEGF pathway as an anti-cancer therapy was demonstrated by the phase III trial of the anti-VEGF monoclonal antibody bevacizumab versus placebo in combination with chemotherapy for metastatic colorectal cancer. In this trial the addition of bevacizumab to chemotherapy showed a statistically significant improvement in overall survival for these subjects (11). Since this trial, the addition of bevacizumab to chemotherapy has been shown to be beneficial in non-small cell lung cancer subjects and metastatic breast cancer subjects (9, 12).

Integrins have been shown to be essential components of angiogenesis. One of the best-characterized integrins in tumor-induced angiogenesis is αvβ3. Angiogenesis dramatically up-regulates integrin αvβ3 expression by endothelial cells (13). Integrin αvβ3 has been linked to cell migration and invasion (14), and cell survival (15). Inhibition of αvβ3 results in apoptosis of endothelial cells (16) and inhibition of microvascular network formation (17). The signaling pathways activated by αvβ3 and VEGF act synergistically in the formation of microvascular networks (17). Both αvβ3 and VEGF activate Src, Ras, PI3K, and Erk cascades (18). CNTO 95 is a fully humanized monoclonal antibody that blocks integrin αvβ3 with high affinity.

The combination of different targeted therapies has the potential of providing a more complete inhibition of angiogenesis. It is our hypothesis that the combination of CNTO 95 and bevacizumab will be a safe and potentially efficacious anti-angiogenesis strategy for the treatment of adult solid tumors. This combination may have utility directly or may prove useful when subsequently combined with other anti-angiogenic agents or standard chemotherapy regimens. We also hypothesize that our clinical dermal wound angiogenesis assay will help quantify and characterize the anti-angiogenic contribution of each agent in this combination.

Bevacizumab (Avastin) is a humanized monoclonal antibody to VEGF. VEGF is known to play a pivotal role in tumor angiogenesis and is a significant mitogenic stimulus for arterial, venous and lymphatic endothelial cells. The addition of bevacizumab to chemotherapy has been shown to increase overall response rate, duration of response and survival for patients with metastatic colon cancer (4) and is beneficial in first line non-small cell lung cancer and metastatic breast cancer [1, 2], and second line metastatic colorectal cancer (7). VEGF signals through phosphotidylinositol 3-kinase (PI3K) and Akt as well as through the extracellular regulated kinase (ERK 1/2), a mitogen activated protein kinase (MAPK). VEGF's multiple biologic actions may be mediated by different pathways. Erikkson demonstrated that VEGF induced hyperpermeability was highly dependent on activation of the AKT pathway, while the angiogenic effect was largely unaffected by blocking this pathway and likely depended on ERK activation [3].

CNTO 95 is a fully human mAb immunoglobulin G (IgG) of the gamma isotype and kappa light chain that has been shown to have antiangiogenic and antitumor properties. Results of in vitro studies demonstrate that CNTO 95 is an anti-αv integrin antibody that binds and blocks integrin ανβ3 with high affinity. CNTO 95 has also been shown to bind to integrins ανβ1, ανβ5, and ανβ6. No cross-reactivity of CNTO 95 to glycoprotein IIb/IIIa, ανβ1 or platelets has been observed. By binding and blocking the ανβ3 and ανβ5 integrins, CNTO 95 can inhibit cell adhesion, migration, proliferation, and invasion of both tumor and endothelial cells in vitro. It is known that CNTO 95 binds to other αν integrins. However, the clinical implications of binding to these integrins are unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of advanced solid tumor refractory to standard therapy or for whom there is no standard therapy. Disease must be measurable by RECIST criteria.
2. Age ≥ 18 years.
3. Karnofsky performance status ≥ 70%.
4. Life expectancy of at least 3 months.
5. Patients must have adequate organ and marrow function as defined below:

   Absolute neutrophil count ≥ 1,500/μl Platelets ≥ 100,000/μl Total bilirubin ≤ 1.5 X upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 2.5 X ULN, ≤ 5 X ULN if known hepatic metastases Creatinine clearance ≥ 50 mL/min/m2 for patients with creatinine levels (by Cockroft-Gault equation or 24 hour urine) Hemoglobin > 9 g/dL Continuation of erythropoietin products is permitted. Hemoglobin must be stable above 9 g/dL for at least 2 weeks without blood transfusion to maintain hemoglobin level.

   Calcium (corrected for albumin) > 8.7 mg/dL
6. The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be embryo- and feto- toxic. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician and study PI immediately. Subjects who are pregnant and/or lactating are excluded from this study.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subjects who have had radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for cancer within the 28 days prior to day 1 of study treatment. Subjects must not have had major surgery within the 28 days prior to study treatment day 1 or minor surgical procedures within the 7 days prior to study treatment day 1.
2. Subjects who have received any other investigational agents within the 28 days prior to day 1 of the study.
3. Subjects with known CNS metastases, centrally located non-small cell lung cancer (regardless of histologic sub-type), non-small cell lung cancer of squamous histology, and/or history of hemoptysis (> ½ tsp BRB).
4. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg). Initiation of antihypertensive is permitted provided adequate control is documented 3 times over at least 1 week before starting treatment.
5. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
6. Evidence of bleeding diathesis or coagulopathy. Subjects on therapeutic anticoagulation may be enrolled provided that they have been clinically stable on anti-coagulation for at least 2 weeks.
7. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of study treatment (56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study
8. Core biopsy or other minor surgical procedure excluding study-related procedures or placement of a vascular access device, within 7 days prior to expected start of treatment.
9. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
10. Serious, non-healing wound, ulcer, or bone fracture
11. Proteinuria at screening as demonstrated by either urine protein:creatinine (UPC) ratio ≥ 1.0 or 24hr collection >1g/24hr at screening
12. Any prior history of hypertensive crisis or hypertensive encephalopathy
13. New York Heart Association (NYHA) Grade II or greater congestive heart failure
14. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to day 1 of study treatment
15. History of stroke or transient ischemic attack within 6 months prior to day 1 of study treatment
16. History of intolerance or hypersensitivity to prior treatment with bevacizumab or CNTO 95. Prior treatment with these agents is permitted, as long as prior treatment was with only one agent at a time (ie - subjects may not have previously received bevacizumab and CNTO 95 together).
17. Chronic treatment with systemic steroids or another immunosuppressive agent, though steroids may be used on an as-needed basis - ie - for treatment of nausea. Treatment with megace or low dose glucocorticoids is permitted for treatment of anorexia.
18. Other known concurrent severe and/or uncontrolled medical disease which could compromise safety of treatment as so judged by treating physician (i.e., severely impaired lung function, uncontrolled diabetes (history of consistent blood glucose readings above 300 mg/dL or less than 50 mg/dL), uncontrolled hypertension (greater than 150/100), severe infection, severe malnutrition, ventricular arrhythmias active ischemic heart disease, known active vasculitis of any cause, tumor invasion of any major blood vessel, chronic liver or renal disease, active upper GI tract ulceration)
19. A known history of HIV seropositivity,hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.
20. Subjects with an active, bleeding diathesis or on oral anti-vitamin K medication (except coumadin). No history of active GI bleeding or other major bleeding within previous 6 months.
21. Subjects unwilling to or unable to comply with the protocol
22. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety or compliance with study requirements or may interfere with the interpretation of the results.
23. Known history of anaphylaxis allergic reactions to human Ig therapy or polysorbate 80 (components of CNTO 95).
24. Known history of uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To define a recommended phase II dose for the combination of CNTO 95 plus bevacizumab in subjects with advanced solid tumors. | Every cycle (21 days)
To evaluate dose limiting as well as non-dose limiting toxicities of this combination. | Every cycle (21 days)

SECONDARY OUTCOMES:
To explore the effect of the combination versus each agent individually on dermal wound angiogenesis in a skin biopsy, the clinical activity of this combination, and the association between blood- and urine-based biomarkers and clinical outcome. | Every cycle (21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States